CLINICAL TRIAL: NCT01728909
Title: The Effects of Intranasal Oxytocin on Social Cognition and Social Approach Behaviors in Opioid-dependent Patients
Brief Title: Methadone Oxytocin Option
Acronym: MOO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Woolley, Assistant Professor in Residence, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-07691
Record Dates: First submitted 2012-11-07; First posted 2012-11-20 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Substance Abuse; Opioid Dependence; Methadone Treatment
Keywords: Oxytocin; Syntocinon; Social Cognition; Social Approach Behaviors
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): 40 IU Oxytocin
  Interventions: Drug: Oxytocin
- Saline Nasal Spray (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Saline Nasal Spray

INTERVENTIONS:
Drug: Oxytocin — 40 IU of the oxytocin will be administered intranasally for a one time dose at the beginning of the visit.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Saline Nasal Spray — 40 IU of the saline nasal spray will be administered once at the beginning of the visit.
  Other Names: Placebo
  Arms: Saline Nasal Spray

SUMMARY:
The purpose of the study is to examine the effects of intranasal oxytocin administration on social cognition in patients receiving methadone maintenance treatment (MMT), examine the effects of intranasal oxytocin administration on opioid craving and on the subjective effects of methadone, and examine the effects of intranasal oxytocin administration on implicit preferences for drug-related and social stimuli in patients receiving MMT.

Hypothesis 1: Patients will perform better on measures of social cognition (including affect recognition and recognition of sarcasm) after administration of oxytocin compared with placebo.

Hypothesis 2: Patients will demonstrate lower craving for opioids and greater subjective effects of methadone after administration of oxytocin compared with placebo.

Hypothesis 3: Patients will demonstrate increased implicit preferences for social stimuli and decreased implicit preferences for drug related stimuli after administration of oxytocin compared with placebo.

ELIGIBILITY:
Inclusion Criteria for patients:

* Primary diagnosis of opioid dependence according to DSM-IV TR
* Opioid of choice be either heroin or oral opioid analgesics
* Currently be on stable dose of methadone with no dose change in the last 14 days

Inclusion Criteria for healthy volunteers

-No diagnosis of mental disorder according to DSM-IV TR

Exclusion Criteria for patients and healthy volunteers:

* Epilepsy
* Current illicit drug use (within the past one month)
* Current sever depression with suicidal thoughts and/or actions
* Addiction to alcohol or drugs other than opiates, caffeine, or nicotine
* Psychotic illness
* Bipolar disorder
* Brain trauma
* Severe Neuropsychological disorder
* Kidney Disease (i.e., kidney stones, recurrent bladder infections, or known kidney failure)
* Sensitivity to preservatives (in particular E216, E218, and chlorobutanol hemihydrate)
* Nasal obstruction, discharge, or bleeding
* Cardiovascular problems (e.g., heart disease, history of heart attacks), high blood pressure (hypertension)
* Habitually drink large volumes of water

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Computerized Social Cognition Tasks | Participants will complete 2 days of the study. These 2 days will be at least a week apart.
  Participants will undergo computer tasks that measure social cognition, which include the TASIT, RMET, and the IAT. The TASIT measures the awareness of social inference, the RMET measures the ability to guess the emotions of others, and the IAT measures implicit associations.

SECONDARY OUTCOMES:
Craving Questionnaires | Participants will complete 2 days of the study. These 2 days will be at least a week apart.
  Participants are asked to rate their current symptoms and current craving levels and for different substances.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, MD, PhD, Principal Investigator — University of California San Francisco, San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Woolley JD, Arcuni PA, Stauffer CS, Fulford D, Carson DS, Batki S, Vinogradov S. The effects of intranasal oxytocin in opioid-dependent individuals and healthy control subjects: a pilot study. Psychopharmacology (Berl). 2016 Jul;233(13):2571-80. doi: 10.1007/s00213-016-4308-8. Epub 2016 May 3. PMID 27137199